CLINICAL TRIAL: NCT00092573
Title: Evaluation of the Efficacy and Safety of Fenofibrate and Ezetimibe Coadministration in Patients With Mixed Hyperlipidemia
Brief Title: Study of Ezetimibe and Fenofibrate in Patients With Mixed Hyperlipidemia (0653-036)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0653-036 Extension; 2004_036
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Hypertriglyceridemia
Keywords: Mixed hyperlipidemia (high cholesterol and high triglycerides)
MeSH Terms: conditions — Hypercholesterolemia; Hypertriglyceridemia; Hyperlipoproteinemia Type II | interventions — Ezetimibe

INTERVENTIONS:
Drug: MK0653, ezetimibe
Drug: Comparator: fenofibrate monotherapy

SUMMARY:
The purpose of this study is to assess the cholesterol lowering safety and effectiveness of two investigational drugs in patients with mixed hyperlipidemia (high cholesterol and high triglycerides).

DETAILED DESCRIPTION:
The duration of treatment is 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* High cholesterol and high triglycerides

Exclusion Criteria:

* Patient has a condition which, in the opinion of the investigator, might pose a risk to the patient, interfere with participation in the study, or does not meet the additional criteria as required by the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2003-04; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Tolerability

SECONDARY OUTCOMES:
Plasma LDL-C, HDL-C and triglycerides after 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Farnier M, Freeman MW, Macdonell G, Perevozskaya I, Davies MJ, Mitchel YB, Gumbiner B; Ezetimibe Study Group. Efficacy and safety of the coadministration of ezetimibe with fenofibrate in patients with mixed hyperlipidaemia. Eur Heart J. 2005 May;26(9):897-905. doi: 10.1093/eurheartj/ehi231. Epub 2005 Mar 21. PMID 15781429
- [Background] McKenney JM, Farnier M, Lo KW, Bays HE, Perevozkaya I, Carlson G, Davies MJ, Mitchel YB, Gumbiner B. Safety and efficacy of long-term co-administration of fenofibrate and ezetimibe in patients with mixed hyperlipidemia. J Am Coll Cardiol. 2006 Apr 18;47(8):1584-7. doi: 10.1016/j.jacc.2005.11.072. Epub 2006 Mar 30. PMID 16630994
- [Background] Tribble DL, Farnier M, Macdonell G, Perevozskaya I, Davies MJ, Gumbiner B, Musliner TA. Effects of fenofibrate and ezetimibe, both as monotherapy and in coadministration, on cholesterol mass within lipoprotein subfractions and low-density lipoprotein peak particle size in patients with mixed hyperlipidemia. Metabolism. 2008 Jun;57(6):796-801. doi: 10.1016/j.metabol.2008.01.026. PMID 18502262
- [Derived] Farnier M, Dong Q, Shah A, Johnson-Levonas AO, Brudi P. Low incidence of paradoxical reductions in HDL-C levels in dyslipidemic patients treated with fenofibrate alone or in combination with ezetimibe or ezetimibe/simvastatin. Lipids Health Dis. 2011 Nov 16;10:212. doi: 10.1186/1476-511X-10-212. PMID 22087637